CLINICAL TRIAL: NCT06789744
Title: Enhanced Recovery After Urologic Surgery: a Prospective Observational Study Comparing Regional with Conventional Anesthetic Techniques
Brief Title: Enhanced Recovery After Urologic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaguang Duan (Other)
Responsible Party: Sponsor-Investigator, Xiaguang Duan, Deputy Chief of Anesthesiology, Inner Mongolia Baogang Hospital
Organization: Inner Mongolia Baogang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-MER-315
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Circumcision; Hydrocelectomy; Hernia; Renal Cyst; Prostate
MeSH Terms: conditions — Hernia | interventions — Anesthesia, General; Analgesia, Epidural; Ropivacaine; Analgesia, Patient-Controlled; Passive Cutaneous Anaphylaxis; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- EA group (Experimental): For epidural analgesia, an initial bolus of 5-15 mL of 0.5% ropivacaine will be administered, followed by a continuous infusion of 0.2% ropivacaine at a rate of 3-10 mL/hour. In pediatric patients, the initial bolus will consist of 0.2% ropivacaine at a dose of 0.5-1 mg/kg, not to exceed 2-2.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hour.
  Interventions: Procedure: Epidural Analgesia( 0.2% ropivacaine)
- PVB group (Experimental): For paravertebral blocks, patients will be positioned either sitting or in the lateral decubitus position to fully expose the target area of the spine. The spinous process of the target vertebra will be palpated, and the puncture site identified. Using ultrasound guidance, the paravertebral space will be located. After standard skin preparation, a blunt needle will be advanced perpendicular to the skin. Once the needle tip contacts the transverse process, it will be withdrawn 1-2 mm, and then slightly angled caudally to pass through the paravertebral ligament and enter the paravertebral space. After negative aspiration for blood or cerebrospinal fluid, a 5 mL test dose of local anesthetic will be slowly injected, and the patient observed for adverse effects. If none are noted, an additional 5 mL of local anesthetic will be injected. The local anesthetic solution will be either liposomal bupivacaine (266 mg diluted to 20 mL) or 0.2% ropivacaine.
  Interventions: Device: General Anesthesia (GA); Device: Paravertebral block ( liposomal bupivacaine 133 mg or 0.2% ropivacaine)
- TAP group (Experimental): For TAP blocks, patients will be positioned supine with the abdomen exposed. Following standard skin preparation, a needle will be advanced perpendicular to the skin using ultrasound guidance, through the external oblique and internal oblique muscles to reach the fascial plane between the transversus abdominis and internal oblique muscles. After negative aspiration for blood, a 5 mL test dose of local anesthetic will be slowly injected, and the patient observed for adverse effects. If none are noted, an additional 10 mL of local anesthetic will be injected. The local anesthetic solution will be either liposomal bupivacaine (266 mg diluted to 20 mL) or 0.2% ropivacaine.
  Interventions: Device: General Anesthesia (GA); Device: Transversus Abdominis Plane Block (TAP Block)( liposomal bupivacaine 133 mg or 0.2% ropivacaine)
- IM group (Experimental): For intrathecal analgesia, adults will receive 0.1-0.2 mg of morphine intrathecally. For pediatric patients, the dose of intrathecal morphine will be 5-10 mcg/kg.
  Interventions: Procedure: Epidural Analgesia( 0.2% ropivacaine); Procedure: Intrathecal Morphine
- PCA group (Active Comparator): For intravenous PCA, a solution of fentanyl 2 mcg/kg will be diluted to a total volume of 100 mL with normal saline. The PCA settings will be as follows: a basal rate of 2 mL/hour, a PCA dose of 2 mL, and a lockout interval of 15 minutes.
  Interventions: Device: General Anesthesia (GA); Drug: Intravenous Patient-Controlled Analgesia (PCA) (fentanyl)

INTERVENTIONS:
Device: General Anesthesia (GA) — Patients will be induced with general anesthesia, consisting of propofol (1.5-2 mg/kg intravenously), rocuronium (1-2 mg/kg intravenously), and fentanyl (1-2 μg/kg intravenously). Anesthesia will be maintained with inhaled sevoflurane or desflurane, adjusted according to BIS values. Remifentanil (0.05-0.2 μg/kg/min) will be administered via continuous infusion, with the infusion rate adjusted to maintain blood pressure and heart rate within ±20% of baseline.
  Following induction, patients will be mechanically ventilated in pressure-regulated volume control (PRVC) mode using an Aestiva anesthesia machine (GE Healthcare, Waukesha, Wisconsin, USA). Ventilator settings will be as follows: tidal volume 6-8 mL/kg, positive end-expiratory pressure 0 cmH2O, inspiratory-to-expiratory ratio 1:2, respiratory rate 16 breaths per minute (BPM), and inspired oxygen concentration of 41%.
  Arms: PCA group; PVB group; TAP group
Procedure: Epidural Analgesia( 0.2% ropivacaine) — For epidural analgesia, an initial bolus of 5-15 mL of 0.5% ropivacaine will be administered, followed by a continuous infusion of 0.2% ropivacaine at a rate of 3-10 mL/hour. In pediatric patients, the initial bolus will consist of 0.2% ropivacaine at a dose of 0.5-1 mg/kg, not to exceed 2-2.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hour.
  Arms: EA group; IM group
Device: Paravertebral block ( liposomal bupivacaine 133 mg or 0.2% ropivacaine) — For paravertebral blocks, patients will be positioned either sitting or in the lateral decubitus position to fully expose the target area of the spine. The spinous process of the target vertebra will be palpated, and the puncture site identified. Using ultrasound guidance, the paravertebral space will be located. After standard skin preparation, a blunt needle will be advanced perpendicular to the skin. Once the needle tip contacts the transverse process, it will be withdrawn 1-2 mm, and then slightly angled caudally to pass through the paravertebral ligament and enter the paravertebral space. After negative aspiration for blood or cerebrospinal fluid, a 5 mL test dose of local anesthetic will be slowly injected, and the patient observed for adverse effects. If none are noted, an additional 5 mL of local anesthetic will be injected. The local anesthetic solution will be either liposomal bupivacaine (266 mg diluted to 20 mL) or 0.2% ropivacaine.
  Arms: PVB group
Device: Transversus Abdominis Plane Block (TAP Block)( liposomal bupivacaine 133 mg or 0.2% ropivacaine) — For TAP blocks, patients will be positioned supine with the abdomen exposed. Following standard skin preparation, a needle will be advanced perpendicular to the skin using ultrasound guidance, through the external oblique and internal oblique muscles to reach the fascial plane between the transversus abdominis and internal oblique muscles. After negative aspiration for blood, a 5 mL test dose of local anesthetic will be slowly injected, and the patient observed for adverse effects. If none are noted, an additional 10 mL of local anesthetic will be injected. The local anesthetic solution will be either liposomal bupivacaine (266 mg diluted to 20 mL) or 0.2% ropivacaine.
  Arms: TAP group
Procedure: Intrathecal Morphine — For intrathecal analgesia, adults will receive 0.1-0.2 mg of morphine intrathecally. For pediatric patients, the dose of intrathecal morphine will be 5-10 mcg/kg.
  Arms: IM group
Drug: Intravenous Patient-Controlled Analgesia (PCA) (fentanyl) — For intravenous PCA, a solution of fentanyl 2 mcg/kg will be diluted to a total volume of 100 mL with normal saline. The PCA settings will be as follows: a basal rate of 2 mL/hour, a PCA dose of 2 mL, and a lockout interval of 15 minutes.
  Arms: PCA group

SUMMARY:
This clinical trial aims to investigate the analgesic efficacy of several perioperative pain management strategies-specifically, epidural analgesia, paravertebral blockade, transversus abdominis plane (TAP) block, intravenous patient-controlled analgesia (PCA), and intrathecal morphine-in patients undergoing a range of urological procedures. These procedures include pediatric circumcision, hydrocelectomy, inguinal hernia repair, renal cyst excision, and transurethral resection of the prostate. The trial will also evaluate the safety profiles of two specific local anesthetics, liposomal bupivacaine and ropivacaine. The primary research question is whether these different analgesic techniques reduce postoperative opioid requirements in patients undergoing urological surgery. A secondary question explores the adverse events associated with the use of liposomal bupivacaine and ropivacaine in this population.

Participants will be:

Urological surgery patients undergoing one of the aforementioned procedures. These participants will be randomized to receive one of the following pain management modalities: epidural analgesia, paravertebral blockade, TAP block, intravenous PCA, or intrathecal morphine. Patient assessments will be conducted in the post-anesthesia care unit (PACU) and at 2, 6, 12, and 24 hours postoperatively. Outcome measures will include: Numeric Rating Scale (NRS) pain scores, total postoperative analgesic consumption, recovery status, patient satisfaction, and time to return of bowel function.

DETAILED DESCRIPTION:
This study is designed as a prospective, randomized, comparative trial, employing a double-blind approach, involving both patients and clinicians, to evaluate the efficacy and non-inferiority of five perioperative analgesic techniques-namely, epidural analgesia, paravertebral blockade, transversus abdominis plane (TAP) block, intravenous patient-controlled analgesia (PCA), and intrathecal morphine-in patients undergoing urological surgery. This study, which is being conducted at Baogang Hospital in Inner Mongolia, was approved by the Medical Ethics Committee of Baogang Hospital, Inner Mongolia, and adheres to the principles of the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) guidelines. All participants provided informed consent voluntarily prior to enrollment.

A total of 150 patients, categorized as American Society of Anesthesiologists (ASA) physical status I-III and of any age, scheduled for urological surgery between February and May 2025, will be enrolled in this study. These patients will be randomized into one of five treatment groups, each comprising 30 participants. The treatment groups will receive one of the following analgesic interventions: epidural analgesia, paravertebral blockade, transversus abdominis plane (TAP) block, intravenous patient-controlled analgesia (PCA), or intrathecal morphine.

Randomization and Blinding：This study employed block randomization to generate the random allocation sequence. A block size of 6 was set, and the random sequence was generated using dedicated software (the blockrand package in R version 4.3.2). The allocation of the random sequence was performed by an independent third party, and allocation concealment was implemented using sequentially numbered, sealed, opaque envelopes. The research team remained blinded throughout the randomization process and was not involved in the generation or allocation of the random sequence.

Intervention：Upon arrival in the operating room, patients will undergo standard monitoring, including pulse oximetry (SpO2), electrocardiography (ECG), bispectral index (BIS), and non-invasive blood pressure measurement. Patients in the intravenous patient-controlled analgesia (PCA) group will receive intravenous fluid infusion. Patients in the intrathecal morphine group will undergo intrathecal injection of morphine. For patients in the epidural analgesia group, an epidural catheter will be placed following epidural puncture. Patients in the paravertebral blockade group will receive a paravertebral block, and those in the transversus abdominis plane (TAP) block group will receive a TAP block. Ultrasound guidance will be used for the paravertebral and TAP blocks with a SonoSite Edge II system (Fujifilm SonoSite, Bothell, WA, USA) and a linear 13-6 MHz ultrasound probe (HFL50x; Fujifilm SonoSite, Bothell, WA, USA). All participating anesthesiologists will have received prior training in the administration of epidural analgesia, paravertebral blockade, TAP blocks, intravenous PCA, and intrathecal morphine.

Following the aforementioned regional analgesic techniques (except for the epidural group), patients will be induced with general anesthesia, consisting of propofol (1.5-2 mg/kg intravenously), rocuronium (1-2 mg/kg intravenously), and fentanyl (1-2 μg/kg intravenously). Anesthesia will be maintained with inhaled sevoflurane or desflurane, adjusted according to BIS values. Remifentanil (0.05-0.2 μg/kg/min) will be administered via continuous infusion, with the infusion rate adjusted to maintain blood pressure and heart rate within ±20% of baseline.

Following induction, patients will be mechanically ventilated in pressure-regulated volume control (PRVC) mode using an Aestiva anesthesia machine (GE Healthcare, Waukesha, Wisconsin, USA). Ventilator settings will be as follows: tidal volume 6-8 mL/kg, positive end-expiratory pressure 0 cmH2O, inspiratory-to-expiratory ratio 1:2, respiratory rate 16 breaths per minute (BPM), and inspired oxygen concentration of 41%.

Epidural Analgesia: For epidural analgesia, an initial bolus of 5-15 mL of 0.5% ropivacaine will be administered, followed by a continuous infusion of 0.2% ropivacaine at a rate of 3-10 mL/hour. In pediatric patients, the initial bolus will consist of 0.2% ropivacaine at a dose of 0.5-1 mg/kg, not to exceed 2-2.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hour.

Paravertebral Block (PVB): For paravertebral blocks, patients will be positioned either sitting or in the lateral decubitus position to fully expose the target area of the spine. The spinous process of the target vertebra will be palpated, and the puncture site identified. Using ultrasound guidance, the paravertebral space will be located. After standard skin preparation, a blunt needle will be advanced perpendicular to the skin. Once the needle tip contacts the transverse process, it will be withdrawn 1-2 mm, and then slightly angled caudally to pass through the paravertebral ligament and enter the paravertebral space. After negative aspiration for blood or cerebrospinal fluid, a 5 mL test dose of local anesthetic will be slowly injected, and the patient observed for adverse effects. If none are noted, an additional 5 mL of local anesthetic will be injected. The local anesthetic solution will be either liposomal bupivacaine (266 mg diluted to 20 mL) or 0.2% ropivacaine.

Transversus Abdominis Plane Block (TAP Block): For TAP blocks, patients will be positioned supine with the abdomen exposed. Following standard skin preparation, a needle will be advanced perpendicular to the skin using ultrasound guidance, through the external oblique and internal oblique muscles to reach the fascial plane between the transversus abdominis and internal oblique muscles. After negative aspiration for blood, a 5 mL test dose of local anesthetic will be slowly injected, and the patient observed for adverse effects. If none are noted, an additional 10 mL of local anesthetic will be injected. The local anesthetic solution will be either liposomal bupivacaine (266 mg diluted to 20 mL) or 0.2% ropivacaine.

Intrathecal Morphine: For intrathecal analgesia, adults will receive 0.1-0.2 mg of morphine intrathecally. For pediatric patients, the dose of intrathecal morphine will be 5-10 mcg/kg.

Intravenous Patient-Controlled Analgesia (PCA): For intravenous PCA, a solution of fentanyl 2 mcg/kg will be diluted to a total volume of 100 mL with normal saline. The PCA settings will be as follows: a basal rate of 2 mL/hour, a PCA dose of 2 Postoperative follow-up will be conducted in both the post-anesthesia care unit (PACU) and on the hospital ward by two specially trained nurses, who will be blinded to patient allocation. Assessments will be performed either in-person or via telephone at the following time points: in the PACU, and at 2, 6, 12, and 24 hours postoperatively.mL, and a lockout interval of 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* any age.
* American Society of Anesthesiologists (ASA) physical status classification of I-III.
* undergo urological surgery.
* receive one of the following analgesic techniques: epidural analgesia (EA), paravertebral block (PVB), transversus abdominis plane (TAP) block, intravenous patient-controlled analgesia (PCA), or intrathecal morphine.
* provided voluntary informed consent.

Exclusion Criteria:

* a bleeding disorder or coagulopathy.
* infection at the intended puncture site or systemic infection.
* a known allergy to local anesthetics.
* spinal deformity or spinal injury.
* a psychiatric disorder that could impair their ability to cooperate with the study protocol.
* pregnant or breastfeeding.
* severe cardiovascular or pulmonary dysfunction.
* chronic opioid use (defined as >1 month) at high doses.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale(NRS) | At baseline (before therapy), at 2 hours post-treatment, at 6 hours post-treatment, at 12 hours post-treatment, and at 24 hours post-treatment.
  The NRS, Numerical Rating Scale, is a rating system from 0 to 10, where 0 represents "no pain" and 10 represents the worst possible pain.

SECONDARY OUTCOMES:
Total Analgesic Consumption | From surgery to 24 hours post-surgery (cumulative consumption). Hourly consumption will be recorded for the first 24 hours to assess temporal patterns of analgesic use.
  Total consumption of analgesics (opioids and non-opioids) will be recorded in milligrams or milliliters (or equivalent doses) during the study period. This includes:Intravenous analgesics (e.g., fentanyl in PCA), Oral analgesics (e.g., acetaminophen, ibuprofen), Rescue analgesics administered as needed.
Patient Satisfaction Score | At 24 hours post-surgery.
  Patient satisfaction will be evaluated using a 5-point Likert scale ranging from 1 (very dissatisfied) to 5 (very satisfied). Patients will be asked to rate their overall satisfaction with the pain management they received.
Time to First Flatus or Bowel Movement | From the end of surgery up to 24 hours.
  Time in hours from the end of surgery to the first passage of flatus or bowel movement, indicating the return of bowel function.
Occurrence of Adverse Events | At 24 hours after surgery
  Record all adverse events related to the interventions, including but not limited to: Nausea and vomiting, Pruritus (itching), Urinary retention, Respiratory depression, Local anesthetic toxicity (e.g., seizures, cardiac dysrhythmias), Hematoma at the injection site, Infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2026-January 2031
Access Criteria: A proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed.